CLINICAL TRIAL: NCT06908161
Title: A Novel Approach for Capturing Real-world Functional Assessment Outcomes in Participants With a Vision Impairment
Brief Title: Functional Assessments in Vision Impairment
Status: Not yet recruiting | Type: Observational
Sponsor: Center for Eye Research Australia (Other)
Responsible Party: Sponsor
Other Study IDs: 24/1642H
Record Dates: First submitted 2025-03-20; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa (RP); Diabetic Retinopathy (DR); Age Related Macular Degeneration (AMD); Glaucoma; Retinal Dystrophy
MeSH Terms: conditions — Retinitis Pigmentosa; Diabetic Retinopathy; Macular Degeneration; Glaucoma; Retinal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the research project is to validate the use of a novel functional assessment tool designed to document how participants with a vision impairment complete activities of daily living in a real world environment.

DETAILED DESCRIPTION:
There is currently no multisensory tool to assess functional vision in people with a vision impairment. This study is designed to capture and assess the reliability and validity of a novel tool developed by multi-disciplinary experts in ophthalmology, optometry, orthoptics, orientation and mobility (O&M) specialists, and people with lived experience of low vision. The tool is designed to be used in both clinical and in interventional clinical trial setting, to provide functional vision assessment measures within real-world outcomes. The development of this tool is at a critical junction in time where a range, of interventions are being developed for people with low vision including bionic eyes, and gene and cell therapies. The FDA requires trials to show real world functional outcomes in addition to traditional endpoints, hence a tool like the ATOMM may have wide use and implications. This study will recruit participants with varying levels of vision impairment to assess the reliability of the ATOMM.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide signed informed consent.
2. Be available for study visits.
3. Willing to comply with study assessments.
4. In good general health and ambulant.
5. Aged over 18 years of age.
6. Have a vision impairment caused by any ocular condition which affects independent mobility.
7. Agree to allow the research team into their home and local environments.
8. Participate in assessments in public settings

Exclusion Criteria:

1. Significant co-morbidities which prohibit involvement in study visits.
2. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
3. Cognitive deficiencies, including dementia or progressive neurological disease.
4. Have a psychiatric condition that, in the investigator's opinion, precludes compliance with the protocol including past or present psychoses and bipolar disorder.
5. Deafness or significant hearing loss.
6. Inability to converse in English.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Centre for Eye Research Australia (CERA) databases will be utilised to identify potential participants. CERA, Cerulea Clinical Trials and the University of Melbourne (UOM) will communicate about the study via social media channels (Facebook, LinkedIn, Twitter), public presentations made by research staff and the via websites.
  Communication may also be distributed in e-newsletters, (such as CERA's Eye-News, or the UOM's newsletters), or print publication (such as CERA's Visionary or Annual Review), and may also form part of an editorial style article which includes information about inherited retinal diseases, glaucoma, age-related macular degeneration and other eye conditions and their prevalence in Australia and the broader opportunities to take part in clinical research.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating validity and reliability | From enrolment to assessment could range from 2 to 4 weeks.
  Two investigators will attend the local environments of each participant for repeated sessions at least two weeks apart to conduct functional assessments using the ATOMM. The tool contains 3 domains involving 15 pre-determined tasks, each designed to encompass common activities of daily living. An example includes independently navigating around the home. A maximum score of 30 points/domain is achievable on a 7 point Likert scale. The investigators will use intraclass correlation coefficients (ICC) to quantify the interrater agreement between two assessors and test-retest reliability over the three domains across the two sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Penelope J Allen, FRACO, FRACS, Principal Investigator — Center for Eye Research Australia
Locations (1):
- Centre for Eye Research Australia, Melbourne, Victoria, Australia